CLINICAL TRIAL: NCT00251303
Title: An Investigation of the Efficacy in Childhood Obsessive-Compulsive Disorder of Riluzole: An Antiglutamatergic Agent
Brief Title: Riluzole to Treat Child and Adolescent Obsessive-Compulsive Disorder With or Without Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Swedo, M.D., Chief, Pediatrics and Developmental Neuroscience Branch, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050225; 05-M-0225 (Other: NIMH Office of Protocol Services)
Record Dates: First submitted 2005-11-09; First posted 2005-11-09 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Obsessive-Compulsive Disorder; Autism Spectrum Disorder; Autism; Asperger Disorder; Developmental Disorder
Keywords: Clinical Trial; Glutamate Antagonist; Pediatrics; Basal Ganglia; Neuropsychological; Obsessive Compulsive Disorder; OCD; Riluzole; Rilutek
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Developmental Disabilities | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- riluzole (Experimental): Active drug put into 10-mg capsule form,,prepared by Clinical Center Pharmacy. Dose up to 120 mg daily, divided. Brand name Rilutek.
  Interventions: Drug: Riluzole
- placebo (Placebo Comparator): Placebo Capsules designed to mimic active drug capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — Active drug put into 10-mg capsules by NIH Clinical Center Pharmacy. Matched placebo capsules were also prepared by NIH Clinical Center Pharmacy. Dose up to 120 mg daily, divided into bid dosages.
  Other Names: Rilutek
  Arms: riluzole
Drug: Placebo — Capsules matched active drug in appearance.
  Arms: placebo

SUMMARY:
This study will examine the effectiveness of riluzole for treating Obsessive-Compulsive Disorder in Youth, Including those with Autism Spectrum Disorders.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic psychiatric disorder characterized by the presence of intrusive and unwanted obsessional thoughts and images and of compulsive behaviors. Its presentation during childhood is similar to that seen in adulthood, except that children sometimes lack insight into the senselessness of the thoughts and behaviors. Although many patients benefit from treatment with selective serotonin reuptake inhibitors (SSRIs), a significant proportion have limited or no response to these medications. Cognitive behavioral therapy (CBT) may also be effective for OCD, alone or in combination with SSRIs, but there is a shortage of qualified therapists, and many patients and families cannot participate effectively in the therapy.

There is a pressing need, then, for the development of alternative, novel treatments for pediatric OCD. Neuropsychological and neuroimaging data suggest that OCD may arise from dysfunction of orbitofronto-striato-thalamocortical circuitry. Glutamate plays a crucial role in the regulation of excitatory activity within this circuit and may be involved in the etiopathogenesis of OCD. If so, then agents which reduce glutamatergic neurotransmission may provide unique antiobsessional benefits. Riluzole is a medication that reduces glutamatergic activity. A small open-label trial suggested that it might reduce OCD severity among children and adolescents.

The investigation will enroll up to 80 pediatric subjects with OCD including some who have both autistic spectrum disorder (ASD) and OCD. The subjects will participate in a double-blind, placebo-controlled 12-week trial of riluzole as a sole agent or as an augmentation to their currently inadequate therapy. Following the double-blind portion of the trial, subjects may receive three months of open-label treatment with riluzole, if it is clinically indicated. All subjects will be followed at regular intervals until one year from baseline.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

1. Male or female subjects, 7 to 17 years of age.
2. Male and female subjects of childbearing potential must be using a medically accepted means of contraception or must remain abstinent.
3. Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study. Each legal guardian must consent to study protocol.
4. Subjects must fulfill DSM-IV criteria for (OCD) and have a CY-BOCS score of greater than 20. In the double-blind phase, subjects enrolled in the combined OCD and ASD cohort must also meet DSM-IV criteria for Pervasive Developmental Disorder as well as OCD.
5. Each subject already taking medicine must be taking usually effective doses of a medicine demonstrated to be effective in childhood OCD, must have been stable on that dose for at least six weeks, and must have no newly recognized or intolerable adverse effects from that medicine. Subjects who are currently not taking such a medication must have had adequate trial in the past of at least one medicine that has been shown to be effective for the symptoms of childhood OCD, and must have failed to see improvement or must have had intolerable adverse effects from the medicine.
6. Subjects must be able to swallow capsules.

EXCLUSION CRITERIA:

Subjects will be excluded from the study for any of the following reasons:

1. Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder, other psychotic disorder, or other serious unstable psychiatric illness. Medically unstable due to binging, purging, or starvation.
2. Judged clinically to be at risk for suicide (suicidal ideation, severe depression, or other factors). Diagnosis of DSM-IV Major Depressive Disorder is not necessarily an exclusion criterion.
3. Disabling Tic Disorder requiring contraindicated medicines.
4. Male or female subjects who are unwilling to use effective contraception, or female subjects who are pregnant or nursing.
5. Serious unstable illnesses, including gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
6. Renal or hepatic dysfunction that would interfere with excretion or metabolism of riluzole as evidenced by increase above upper limits of normal for BUN/creatinine, or more than two-fold elevation above upper limits of normal of serum transaminases (ALT/SGPT, AST/SGOT), gamma glutamate (GGT), or bilirubin.
7. Documented history of hypersensitivity or intolerance to riluzole.
8. DSM-IV Substance Abuse Disorder within the past 90 days or Substance Dependence Disorder within the past 5 years, or any use of tobacco.
9. Taking contraindicated drugs.
10. Unable to swallow capsules.
11. In addition, patients will not receive cognitive-behavior therapy during the period of the study.
12. Abnormal EEG unless evaluated by a neurologist and approved by that specialist for this protocol.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2005-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, MD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sasso DA, Kalanithi PS, Trueblood KV, Pittenger C, Kelmendi B, Wayslink S, Malison RT, Krystal JH, Coric V. Beneficial effects of the glutamate-modulating agent riluzole on disordered eating and pathological skin-picking behaviors. J Clin Psychopharmacol. 2006 Dec;26(6):685-7. doi: 10.1097/01.jcp.0000245567.29531.d6. No abstract available. PMID 17110840
- [Background] Zarate CA Jr, Quiroz JA, Singh JB, Denicoff KD, De Jesus G, Luckenbaugh DA, Charney DS, Manji HK. An open-label trial of the glutamate-modulating agent riluzole in combination with lithium for the treatment of bipolar depression. Biol Psychiatry. 2005 Feb 15;57(4):430-2. doi: 10.1016/j.biopsych.2004.11.023. PMID 15705360
- [Background] Bensimon G, Lacomblez L, Meininger V. A controlled trial of riluzole in amyotrophic lateral sclerosis. ALS/Riluzole Study Group. N Engl J Med. 1994 Mar 3;330(9):585-91. doi: 10.1056/NEJM199403033300901. PMID 8302340
- [Background] Coric V, Milanovic S, Wasylink S, Patel P, Malison R, Krystal JH. Beneficial effects of the antiglutamatergic agent riluzole in a patient diagnosed with obsessive-compulsive disorder and major depressive disorder. Psychopharmacology (Berl). 2003 May;167(2):219-20. doi: 10.1007/s00213-003-1396-z. Epub 2003 Mar 26. No abstract available. PMID 12658528
- [Background] McGrath MJ, Campbell KM, Parks CR, Burton FH. Glutamatergic drugs exacerbate symptomatic behavior in a transgenic model of comorbid Tourette's syndrome and obsessive-compulsive disorder. Brain Res. 2000 Sep 15;877(1):23-30. doi: 10.1016/s0006-8993(00)02646-9. PMID 10980239
- [Background] Moore GJ, MacMaster FP, Stewart C, Rosenberg DR. Case study: caudate glutamatergic changes with paroxetine therapy for pediatric obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 1998 Jun;37(6):663-7. doi: 10.1097/00004583-199806000-00017. PMID 9628087
- [Background] Rosenberg DR, MacMaster FP, Keshavan MS, Fitzgerald KD, Stewart CM, Moore GJ. Decrease in caudate glutamatergic concentrations in pediatric obsessive-compulsive disorder patients taking paroxetine. J Am Acad Child Adolesc Psychiatry. 2000 Sep;39(9):1096-103. doi: 10.1097/00004583-200009000-00008. PMID 10986805
- [Background] Coric V, Taskiran S, Pittenger C, Wasylink S, Mathalon DH, Valentine G, Saksa J, Wu YT, Gueorguieva R, Sanacora G, Malison RT, Krystal JH. Riluzole augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. Biol Psychiatry. 2005 Sep 1;58(5):424-8. doi: 10.1016/j.biopsych.2005.04.043. PMID 15993857
- [Background] Russman BS, Iannaccone ST, Samaha FJ. A phase 1 trial of riluzole in spinal muscular atrophy. Arch Neurol. 2003 Nov;60(11):1601-3. doi: 10.1001/archneur.60.11.1601. PMID 14623733
- [Background] Zarate CA Jr, Payne JL, Quiroz J, Sporn J, Denicoff KK, Luckenbaugh D, Charney DS, Manji HK. An open-label trial of riluzole in patients with treatment-resistant major depression. Am J Psychiatry. 2004 Jan;161(1):171-4. doi: 10.1176/appi.ajp.161.1.171. PMID 14702270
- [Result] Grant PJ, Joseph LA, Farmer CA, Luckenbaugh DA, Lougee LC, Zarate CA Jr, Swedo SE. 12-week, placebo-controlled trial of add-on riluzole in the treatment of childhood-onset obsessive-compulsive disorder. Neuropsychopharmacology. 2014 May;39(6):1453-9. doi: 10.1038/npp.2013.343. Epub 2013 Dec 19. PMID 24356715
- [Derived] Grant P, Lougee L, Hirschtritt M, Swedo SE. An open-label trial of riluzole, a glutamate antagonist, in children with treatment-resistant obsessive-compulsive disorder. J Child Adolesc Psychopharmacol. 2007 Dec;17(6):761-7. doi: 10.1089/cap.2007.0021. PMID 18315448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects had to be symptomatic for at least 6 weeks, with a score of at least 20 CY-BOCS; had to have had at least one standard-of-care treatment for childhood OCD for adequate periods of time; had to have been stable for at least 6 weeks on any medicine; had to meet entrance criteria at a screening and 2 weeks later.
Groups:
- Riluzole: Riluzole was titrated upward to at least 100 mg of active drug. If adverse effects are noted, dose titration was slowed, stopped, or reversed, or the drug was discontinued. Maximum permitted dose of riluzole was 120 mg/day.
- Placebo: Placebo capsules were prepared by NIH Clinical Center Pharmacy to appear identical to active drug capsules. Dose was titrated upward as if active drug. Follow-up and laboratory studies were identical for active drug and placebo arms.
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 30 (78 subjects signed any consent. 60 started drug (30 riluzole & 30 placebo).) | 30
Completed | 22 | 29
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Population: These data apply only to double-blind phase.
Groups:
- Riluzole: In a 12-weeks long double-blind phase, the clinicians and subjects and their guardians were blind to active drug or placebo. There were approx. twice monthly in-person or telephone contacts.
  Riluzole was titrated upward to at least 100 mg of active drug. If adverse effects are noted, dose titration was slowed, stopped, or reversed, or the drug was discontinued. Maximum permitted dose of riluzole was 120 mg/day. At the end of the 12 weeks study period, subjects and their families could elect to take open-label riluzole.Since neither subjects nor investigators knew whether subjects had been receiving active drug,the open-label administration was also titrated. Laboratory assays were obtained at 2, 4, 8, and 12 weeks after starting the open-label riluzole, as they had been during double-blind. Subsequently, testing was less frequent.
- Placebo: Placebo capsules were prepared by NIH Clinical Center Pharmacy to appear identical to active drug capsules. Dose was titrated upward as if active drug. Follow-up and laboratory studies were identical for active drug and placebo arms. At the end of the double-blind phase, subjects could elect to take open-label drug, which was titrated upward to the maximum dose, 100 mg daily.
  Study blind was not broken for subjects or investigators until the final subject had completed the double-blind phase of the study.
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.78 (2.10) | 14.17 (2.58) | 14.47 (2.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Much/Very Much Improved on Clinical Global Impressions - Improvement Score (CGI-I)
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 29
participants | 3 | 4
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority or Other; p = 0.959, Chi-squared

2. Primary Outcome: Children's Yale-Brown Obsessive-Compulsive Scale Scores (CY-BOCS)
Description: CY-BOCS is a 0-40 point scale of obsessive-compulsive symptom severity, higher number indicates more severe obsessive-compulsive symptoms. Comparison of 12 weeks scores for placebo and riluzole groups.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 29
units on a scale | 21.72 (6.43) | 23.30 (4.64)

ADVERSE EVENTS:
Time Frame: 12 weeks double-blind period.
Arm/Group | Riluzole | Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 27/30 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=30) | Placebo (N=30)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Riluzole (N=30) | Placebo (N=30)
chest pain, hypotension, Tachycardia, EKG abnormality, and other cardiovascular (Cardiac disorders) | 8 (11) | 5 (5)
earache, poor hearing, Tinnitus, and ear other (Ear and labyrinth disorders) | 13 (17) | 11 (13)
eye irritation, blurred vision, eye other (Eye disorders) | 6 (9) | 8 (10)
fever (Infections and infestations) | 6 (6) | 7 (7)
Accidental Injury (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Muscle Bone joint pain, Dyskinesia, Muscle Rigidity, and Musclualrsketetal other (Musculoskeletal and connective tissue disorders) | 14 (14) | 12 (15)
Mouth Ulcer, Dry mouth, sore tongue, gum problems, Dental problems, and mouth other (Gastrointestinal disorders) | 11 (18) | 13 (19)
Stomach or abdominal discomfort, nausea, vomitting, diarrhea, constipation, stool discoloration (Gastrointestinal disorders) | 18 (37) | 21 (47)
appetite increase/decrease, taste abnormality, increased thirst, and gastrointestinal other (Gastrointestinal disorders) | 12 (23) | 19 (39)
headache, dizziness, akathisia, tremor, tic movements, slurred speech, and confusion (Nervous system disorders) | 23 (46) | 17 (32)
concentration difficulty and memory problems (Nervous system disorders) | 15 (21) | 13 (20)
Painful urination, difficulty urinating, increased frequency, and enuresis (Renal and urinary disorders) | 9 (11) | 13 (15)
Dermatologic Skin Irritation, Sweating, hair problems, and skin other (Skin and subcutaneous tissue disorders) | 20 (25) | 20 (28)
breast pain swelling, discharge from nipples, menstrual irregularity, cramps, premenstral tension (Reproductive system and breast disorders) | 7/8 (7) | 4/8 (8)
genital discomfort, increased/decreased libido and genitourinary other (Reproductive system and breast disorders) | 5 (7) | 2 (3)
nasal congestion, bloody nose, sore throat, difficulty swallowing, and flu upper respitory (Respiratory, thoracic and mediastinal disorders) | 20 (35) | 24 (44)
nose throat other, shortness of breath, wheezing, and coughing (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 15 (26)
medical or surgical procedure (Surgical and medical procedures) | 1 (1) | 3 (3)
tiredness fatigue, increased/decreased motor activity, difficulty falling asleep (Psychiatric disorders) | 22 (36) | 22 (45)
early morning awakening, interrupted sleep, drowsiness sedation, hallucinations, depression, anxiety (Psychiatric disorders) | 24 (62) | 25 (66)
irritability, suicidal ideas, suicidal behavior, agression, and psychological behavior other (Psychiatric disorders) | 21 (35) | 21 (38)
swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Only treatment-refractory subjects were eligible for study participation. This may have decreased treatment response. Further, 98% were taking psychotropic drugs at baseline, which may have reduced between-group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes